CLINICAL TRIAL: NCT04295213
Title: The Effect of a Oligosaccharides Versus a Placebo on Defecation Parameters in Healthy Children With Hard or Lumpy Stools
Brief Title: The Inside Study II: Oligosaccharides Versus Placebo and Hard Stools
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University and Research (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); FrieslandCampina, Amersfoort, The Netherlands (Unknown)
Responsible Party: Principal Investigator, Clara Belzer, Associate Professor, Wageningen University and Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL70820.081.19
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Healthy With Hard and/or Lumpy Stools
Keywords: oligosaccharides
MeSH Terms: interventions — Oligosaccharides

STUDY DESIGN:
Intervention Model Description: Parallel study with two arms of 13 weeks in total per participant
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oligosaccharide group (Experimental): intervention with oligosaccharides, total duration of study is 13 weeks
  Interventions: Other: oligosaccharides
- placebo group (Placebo Comparator): Placebo comparator, total duration of study is 13 weeks
  Interventions: Other: oligosaccharides

INTERVENTIONS:
Other: oligosaccharides — 1 dose a day of oligosaccharides or placebo

SUMMARY:
In the present randomised double blind controlled study, we will study the effects of a oligosaccharides vs a placebo on the change in stool consistency and stool frequency in children with hard or lumpy stools.

DETAILED DESCRIPTION:
Firm, hard or lumpy stools can be problematic for young children and might come as a precursor of functional constipation in childhood. The cause of harder stools in childhood is incompletely understood. But it is likely that harder stools in childhood are linked to among others withholding behaviour of stools and a low fibre intake. As hard stools may precede functional constipation, the aim of the study is to investigate the effect of a prebiotic fiber versus a placebo on defecation parameters in healthy children with hard or lumpy stools. We hypothesize that consumption of a prebiotic fiber results in softer stools.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* aged 1-4 years
* Hard and/or firm stools as scored by a stool questionnaire

Exclusion Criteria:

* Children that meet the Rome IV criteria for functional constipation
* Children who suffer from any other GI complaints, known structural GI abnormalities, or previous GI surgery
* Any condition that would make it unsafe for the child to participate.
* Children with clinically significant cardiac, vascular, liver, pulmonary, psychiatric disorders, severe renal insufficiency, human immunodeficiency virus, acquired immunodeficiency syndrome, hepatitis B or C or known abnormalities of haematology, urinalysis, or blood biochemistry, as checked by the inclusion questionnaire.
* Children who are allergic to cow's milk or fish
* Use of antibiotics or other medicines or food supplements, and breast milkfeeding, which can influence defecation and gut microbiota 4 weeks prior to the study
* Children that participate in another clinical trial

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 196 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Stool consistency | Stool consistency will be measured at different time points during a study period of 13 weeks.
  Change in stool consistency measured by the a stool questionnaire; 5 points stool scale from 1 hard to 5 watery (modified Bristol Stool Form Scale)

SECONDARY OUTCOMES:
Stool frequency in number of cases (%) | These outcome measures will be measured at different time point during a study period of 13 weeks.
  Stool frequency - number of times a child has stools a day as reported in a diary.by a stool questionnaire
Stool consistency in number of cases (%) | These outcome measures will be measured at different time point during a study period of 13 weeks.
  Stool consistency - % of stools in a certain stool scale score as measured via a 5 point stool scale

CONTACTS AND LOCATIONS:
Overall Officials: Clara Belzer, PhD, Principal Investigator — Wageningen University and Research; Marc Benninga, PhD, Principal Investigator — Emma Children's Hospital, UMC Amsterdam
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No